CLINICAL TRIAL: NCT04358198
Title: Usefulness of Artificial Intelligence (AI) for Gastric Intestinal Metaplasia Diagnosis
Brief Title: AI in GIM Diagnosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Principle investigator, King Chulalongkorn Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RP018
Record Dates: First submitted 2020-04-12; First posted 2020-04-24 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: GIM Diagnosis; Artificial Intellegence
MeSH Terms: interventions — Artificial Intelligence

STUDY DESIGN:
Intervention Model Description: The surveillance EGD in patients with GIM will be done as scheduled and then pictures at GIM lesions and normal mucosa was done and sending to AI for learning. Then AI will be used for diagnosing GIM by using pathology as a gold standard
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GIM patient (Experimental): The patients with GIM will be assessed at both GIM and normal mucosa during endoscopy.
  Interventions: Diagnostic Test: Artificial intelligence

INTERVENTIONS:
Diagnostic Test: Artificial intelligence — The AI algorithm based on the convolutional neural network (CNN) will be used for analysis the pictures of gastric intestinal metaplasia and normal mucosa. Then AI will be used as a diagnostic tool for GIM during routine endoscopy by using pathology as a gold standard.

SUMMARY:
This study will use artificial intelligence (AI) for diagnosing gastric intestinal metaplasia.

DETAILED DESCRIPTION:
The patients with previously diagnose gastric intestinal metaplasia (GIM) and have the surveillance gastroscopy will be enrolled. The routine surveillance program will be performed additional to taking photo at both GIM and normal mucosa at least 5 pictures in each. Biopsy will be done to confirm the diagnosis of GIM and normal mucosa. All pictures will be inserted to AI algorithm based on the convolutional neural network (CNN). Then, the AI program will be validated in daily endoscopy compared with pathology. Accuracy, sensitivity and specificity can be calculated by 2x2 table.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years of age
* Able to sign a consent form

Exclusion Criteria:

* History of gastric surgery
* Coagulopathy
* Pregnancy/Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AI for GIM diagnosis | 1 year
  Accuracy, sensitivity, specificity can be calculated by 2x2 table (pathology is a gold standard)

CONTACTS AND LOCATIONS:
Locations (1):
- Rapat Pittayanon, Pathum Wan, Bangkok, Thailand